CLINICAL TRIAL: NCT06185374
Title: Text Messaging to Improve Adherence To Repeat Colonoscopy In The VA: A Pilot Study
Brief Title: Text Messaging to Improve Adherence To Repeat Colonoscopy In a Veterans Affairs (VA) Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23-00583
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Message Intervention (Experimental): Participants in the experimental arm will receive a series of instructional and motivational text messages, which will be sent starting 7-14 days before and until the day of the colonoscopy procedure.
  Interventions: Behavioral: Text Message Instructions/Motivation
- No Intervention (No Intervention): Participants will not receive text messages.

INTERVENTIONS:
Behavioral: Text Message Instructions/Motivation — For instructional messages, earlier messages will remind patients of the colonoscopy appointment and later messages will help patients complete the bowel preparation process in real-time. Motivational messages will be sent along with instructional messages.
  Arms: Text Message Intervention

SUMMARY:
Colorectal cancer is a common but preventable condition, and increasing colorectal cancer screening is one of the most impactful public health contributions in the field of gastroenterology. Text messaging is a simple, cheap, and rapid method to reach patients that may improve adherence to colonoscopy appointments as well as simplify the process of bowel preparation. The purpose of the study is to evaluate the feasibility of a pilot bidirectional text messaging intervention on attendance for screening/surveillance colonoscopy and bowel preparation quality at an urban VA hospital. The goal is to improve adherence to colonoscopy among patients who are due for a repeat colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

• Has previously undergone a colonoscopy and is currently due for a repeat screening or surveillance colonoscopy at the VA.

Exclusion Criteria:

* Patients not due for screening or surveillance colonoscopy. This will be based on 2020 guidelines from the U.S. Multi-Society Task Force on Colorectal Cancer.
* Patients with personal history of colorectal cancer (CRC)/inflammatory bowel disease/ hereditary colon cancer syndrome or family history of hereditary colon cancer syndrome. These criteria will be determined based on ICD9/10 codes or the medical record.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Liang, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York Harbor Health Care System - Department of Veterans Affairs, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: peter.liang@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to peter.liang@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Message Intervention | No Intervention
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Message Intervention | No Intervention | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.95) | 62.76 (6.86) | 63.88 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 23 | 24 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 21 | 18 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 12 | 28
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: National Annie Colonoscopy Survey Score
Description: 7-item assessment of participant satisfaction with the "Annie" text intervention. Items are rated on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). The total score is the sum of responses and ranges from 7 to 35; higher scores indicate greater satisfaction with the intervention.
Time Frame: Day 21 (Up to 7 Days Post-Procedure)
Population: Control patients were not given text messaging intervention, therefore did not participate in the Annie text message survey. All intervention patients were encouraged to complete the survey, and 16 of 25 did.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Text Message Intervention | No Intervention
Number analyzed (Participants) | 16 | 0
Score on a scale | 29.56 (4.16) |

2. Secondary Outcome: Percentage of Participants Who Attend Scheduled Colonoscopy Appointment
Description: Assessed via patient's electronic health record.
Time Frame: Up to Day 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Text Message Intervention | No Intervention
Number analyzed (Participants) | 25 | 25
Percentage of Participants | 96 | 92

3. Secondary Outcome: Percentage of Participants Who Had Adequate Bowel Preparation at Colonoscopy Appointment
Description: Assessed via patient's electronic health record.
Time Frame: Up to Day 14
Measure: Number; unit: percentage of participants
Arm/Group | Text Message Intervention | No Intervention
Number analyzed (Participants) | 24 | 23
percentage of participants | 79 | 91

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Text Message Intervention | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT06185374/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT06185374/ICF_000.pdf